CLINICAL TRIAL: NCT05012358
Title: Genomic Profiling of Mitochondrial Disease - Imaging Analysis for Precise Mitochondrial
Brief Title: Genomic Profiling of Mitochondrial Disease - Imaging Analysis for Precise Mitochondrial Medicine
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Casimir, LLC (Unknown); Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Ralitza Gavrilova, Associate Professor of Medical Genetics and Neurology, College of Medicine, Mayo Clinic
Other Study IDs: 20-002721
Record Dates: First submitted 2021-08-12; First posted 2021-08-19 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Mitochondrial Myopathies; Mitochondrial DNA Mutation; Mitochondrial Diseases; Chronic Progressive External Ophthalmoplegia With Myopathy; Kearns-Sayre Syndrome
Keywords: Mitochondrial DNA deletion
MeSH Terms: conditions — Mitochondrial Myopathies; Mitochondrial Diseases; Kearns-Sayre Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Cohort: no intervention

SUMMARY:
This study is an observational longitudinal study involving the use of MRIs and video recordings taken at home of patients completing basic tasks. Once consent is obtained, subjects will be asked to schedule an appointment with radiology to undergo the listed MRIs of the heart and/or muscle. Subjects will also be given instructions on how to use the video recording app on their personal devices, or study provided device. The subjects will be followed regularly over the course of two years, submitting video recordings of their movements and reporting to Mayo Clinic for MRIs as scheduled.

DETAILED DESCRIPTION:
Mitochondrial myopathy follows a slowly progressive disease course of gradual worsening of muscle weakness and fatigability. Progressive mitochondrial dysfunction is thought to result in structural muscle deterioration (eventually muscle fiber atrophy/necrosis) and underlie these symptoms. Therefore, the study hypothesis is that longitudinal imaging of muscle will capture mitochondrial (using muscle MRS) and structural (using muscle MRI) abnormalities to inform objectively disease progression by capturing structural and biochemical changes in muscle over time.

Conventional multivariate analysis tools such as partial least squares-discriminant analysis (PLS-DA) and principal component analysis (PCA) will be used to assess variables of importance in discrimination of 3 subgroups based on underlying molecular defect (mitochondrial DNA (mtDNA) mutations and deletions, and nuclear gene mutations (nDNA)).

This will be followed by implementation of Collaborative Laboratory Integrated Reports (CLIR) software, a multivariate pattern recognition software that generates post-analytical interpretive tools. This study proposes to quantitatively measure MRS analytes (i.e. lactate, adenosine triphosphate (ATP), etc.) and structural muscle changes by MRI (edema, fat content, etc.). The capability for interactive data analysis would be necessary because of the nature of mitochondrial myopathy (MM) progression. One of the functionalities of CLIR is the creation of post-analytical tools applicable to either diagnosis of one condition - single condition tool; or differential diagnosis between two conditions with overlapping phenotypes (mtDNA deletions, mtDNA mutations, nDNA mutations) - dual scatter plots. The advantages of CLIR are (1) integration of primary markers with all informative permutations of ratios/biomarkers. Ratios calculated between markers not directly related at the biochemical level are particularly helpful to correct for pre-analytical factors and potential analytical bias (2) adjusted for multiple covariates (age, sex) (3) generating individual plots of disease progression.

This study is an observational longitudinal study involving the use of MRIs and video recordings taken at home of patients completing basic tasks. Subjects will be approached at outpatient appointments, or via phone/mail. Once consent is obtained, subjects will be asked to schedule an appointment with radiology to undergo the listed MRIs of the heart and/or muscle. Subjects will also be given instructions on how to use the video recording app on their personal devices, or study provided device. The subjects will be followed regularly over the course of two years, submitting video recordings of their movements and reporting to Mayo Clinic for MRIs as scheduled. Patients may withdraw from the study at any time without repercussion.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed or suspected primary mitochondrial disorder *Suspected mitochondrial disorder would mean that the patient meets clinical criteria and has either biopsy or biochemical testing that supports the diagnosis.

Exclusion Criteria:

* Pregnant, breastfeeding
* Severe cardiac disease who are unable to undergo all the required testing
* Requiring anesthesia for MRIs
* Has severe claustrophobia
* Has implanted devices

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants in the study should have genetic confirmation or muslce biopsy confirmation along with supporting clinical features of mitochondrial disease with weakness in muscle.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Indicators of disease severity and progression - cardiac movement | 2 years
  Establish the prevalence and severity of specific morbid indicators of disease severity through use of echocardiogram
Indicators of disease severity and progression - cardiac function | 2 years
  Establish the prevalence and severity of specific morbid indicators of disease severity through use of magnetic resonance imaging (MRI) of cardiac muscle
Indicators of disease severity and progression - skeletal muscle function | 2 years
  Establish the prevalence and severity of specific morbid indicators of disease severity through use of magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS) of skeletal muscle
Indicators of disease severity and progression - skeletal muscle movement | 2 years
  Establish the prevalence and severity of specific morbid indicators of disease severity through use of video scoring scale during exercise

CONTACTS AND LOCATIONS:
Overall Officials: Ralitza Gavrilova, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No